CLINICAL TRIAL: NCT06516055
Title: A Phase IIa Non-Blinded Study of Safety, Tolerability and Efficacy of S1B-408 in Women With Orgasmic Dysfunction
Brief Title: Study of S1B-408 in Women With Orgasmic Dysfunction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: S1 Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1B-408-2000
Record Dates: First submitted 2024-07-09; First posted 2024-07-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-11

CONDITIONS: Orgasmic Disorder
Keywords: S1B-408; Orgasmic Disorder; Female Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Intervention Model Description: Rating scales and sexual activity log to establish baseline over one month then open-label treatment with dose titration based on results to determine change, with statistical analysis of group differences between month prior to treatment vs treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- S1B-408 (Experimental): One dose of S1B-408 with up-titration of one of its components after one week as needed and tolerated
  Interventions: Drug: S1B-408

INTERVENTIONS:
Drug: S1B-408 — Medication with multiple monoamine activities

SUMMARY:
This is the first clinical trial of S1B-408 in women with sexual dysfunction. A prior 4-week trial in premenopausal women with Hypoactive Sexual Desire Disorder showed that orgasmic function improved with Lorexys (TM). This pilot trial tests for improvement in orgasmic function, safety, and tolerability of a different but related test article.

DETAILED DESCRIPTION:
S1B-408 is a proprietary combination of agents proven safe and effective in other CNS indications. The combination drug is aimed at treating women's sexual dysfunction disorders. Its two components each have pro-sexual effects. However, the efficacy of each when given alone has been limited. Moreover, each component has side effects which, while benign, may limit the drug's utility: activation (agitation, anxiety, insomnia) with one; sedation (somnolence, fatigue, etc) with the other.

The goal of this trial is to show that, when formulated in the proper (fixed) ratio, the combination of these two drugs strengthens their pro-sexual effects for orgasmic dysfunction while mitigating the opposing side effect profiles.

For this pilot study, the goal for exposure is to seek rapid onset of action with minimal dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 60.
2. In a sexual relationship and sexually active within the past month
3. Diagnosis of ICD-10 2023 Orgasmic Dysfunction, secondary or primary. See Investigator's Brochure, section 2, "Medical Need and Diagnosis" for rationale.
4. Orgasmic Dysfunction is the predominant form of sexual dysfunction, is acquired rather than lifelong, and is generalized rather than situational.
5. At screen and baseline visit, scores <8 on the raw score of the FSFI orgasm domain (at least moderate severity)
6. May have depression and/or anxiety if condition is no worse than mild with treatment and if patient will continue the same treatment for the duration of this trial
7. Side effects from any continuing concomitant medications must be stable.
8. Not pregnant or lactating for six months; using contraception that is medically reliable in the investigator's judgment, or (if the investigator finds the patient credibly monogamous) vasectomy of male partner. If hormonal contraception is used, the same medication must have been used for at least 3 months.
9. Gives informed consent for and is willing to undergo all of the scheduled evaluations
10. Prompt for screening and baseline visits, is cooperative, and takes reasonable directions without excessive explanations
11. Her sexual partner is sexually unimpaired (erectile dysfunction allowed only if adequately treated), and available to the subject at least half of the time (in days per week).
12. Agrees to have sexual activity with her partner at least once a week for the duration of her participation in this study.

Exclusion Criteria:

1. Masturbates to orgasm more than once a week.
2. Sexual aversion or sexual pain disorder
3. Chronic conditions that, in the investigator's judgment, are likely to deteriorate within 3 months of screening are not allowed (e.g., gastrointestinal bleeding, uncontrolled diabetes, frequent asthma attacks, uncontrolled Major Depressive disorder, history within the prior 6 months of suicidality or drug abuse; recurrence within the prior year of breast, cervical, uterine, ovarian or other systemic cancer). However, chronic conditions with a relatively stable course are allowed; see Investigator's Brochure, section 2, "Medical Need and Diagnosis" for rationale.
4. Requires CYP3A4, CYP 2B6, or CYP 2D6 strong inhibitor or inducer drugs
5. History of bipolar and/or psychotic disorders and/or takes an antiepileptic/mood stabilizer, antipsychotic, or opioid drug
6. History of severe, serious, or allergic adverse reaction(s) to stimulants or sedatives
7. Drinks >2 alcoholic drinks per day (12-oz beer, 4-oz wine, 1 ½ oz liquor, etc.)
8. History of seizures or use of antiepileptic medication
9. Long QT syndrome (QTc >480 msec), other significant cardiovascular disease
10. moderate or severe dysfunction of the liver (any LFT >3x ULN) or renal dysfunction (BUN > 30 or Cr >2.0)
11. History of blood clots or abnormal bleeding tendencies, including daily use of medications adversely affecting coagulation, e.g., NSAIDs, systemic corticosteroids, or >81 mg aspirin daily.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI): orgasm domain | 7 or 28 day recall
  sum of 3 items on orgasmic frequency, difficulty, and satisfaction, each rated 0 or 1 (worst) to 5 (best)

SECONDARY OUTCOMES:
Changes in Sexual Function Questionnaire (CSFQ): orgasm | 7 day recall
  sum of 3 items on orgasmic frequency, pleasure, and ability, each rated 1 (worst) to 5 (best)
CSFQ total score | "now" or 7 day recall
  sum of 14 items on all aspects of female sexual response, scored from 14 to 70 (best)
FSFI total score | Prior 7 or 28 days
  sum of 19 items on 6 aspects of female sexual response, scored from 4 (worst) to 95 (best)
Female Sexual Distress Scale-Desire/Arousal/Orgasm (FSDS-DAO) items 13, 14, and 15 scores | Prior 7 or 28 days
  3 items on sexual distress re desire, arousal, and orgasm, each scored from 0 to 4 (best)
Sexual Activity Log (SAL), orgasms | 1-7 day recall
  Sexual Activity Log count of orgasms
SAL proportion of sexual activities with orgasm | 1-7 day recall
  Sexual Activity Log count of orgasms over times engaged in sex; best would be 1.0
Sexual Activity Log (SAL) satisfying sexual events | 1-7 day recall
  Count of sexual events that were satisfying
Patient's Global Impression of Change | 4 weeks
  single question rated from 1 (best) to 7 (worst) asking improvement vs none or worsening

OTHER OUTCOMES:
Safety: adverse events | 4-week recall
  All adverse outcomes in clinician's judgment in answer to a question: How do you feel? or in interpreting objective information about the patient
pulse rate | one fourth to one half minute
  number of heart beats per minute effective enough to reach the arm
Blood pressure | one half minute or less
  pressures in mm of mercury when a heartbeat reaches the arm and between heartbeats
Q-T interval | three heartbeats up to the number of heartbeats in 30 seconds
  time in milliseconds between start and end of a contraction of the ventricles of the heart as measured by electrocardiogram (ECG)
Cardiac rate | 1/2 to 1 minute
  Number of contractions of the ventricles of the heart per minute as measured by ECG
Columbia Suicide Severity Rating Scale, 6-item Screening/Triage version (C-SSRS-6) | prior 30 days
  6-item self-rating scale on suicidal ideas, intent and behavior monitored by clinician; "no" rather than "yes" answer to each item is best score
Patient Health Questionnaire-9 Symptom Checklist (PHQ-9) | prior 2 weeks
  9 items on depressive symptoms rated from 0 (best) to 3 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas E Sitchon, B.S., Study Chair — S1 Biopharma, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pyke RE, Clayton AH. Dose-Finding Study of Lorexys for Hypoactive Sexual Desire Disorder in Premenopausal Women. J Sex Med. 2019 Dec;16(12):1885-1894. doi: 10.1016/j.jsxm.2019.09.005. Epub 2019 Oct 31. PMID 31678098